CLINICAL TRIAL: NCT04756687
Title: A Retrospective Analysis in Real World on Lymphocyte Reconstitution After Lymphopenia in Patients Treated by Tecfidera and Description of Management Strategies in France
Brief Title: Real World Analysis on Lymphocyte Reconstitution After Lymphopenia in Participants Treated by Tecfidera
Acronym: Lympho-TEC
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: FR-BGT-11758
Record Dates: First submitted 2021-02-12; First posted 2021-02-16 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting | interventions — Dimethyl Fumarate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: RRMS participants treated with DMF will be identified in the Observatoire Français de la Sclérose en Plaques (OFSEP) database for OFSEP sites.
  Interventions: Drug: Dimethyl fumarate

INTERVENTIONS:
Drug: Dimethyl fumarate — Administered as specified in the treatment arm.

SUMMARY:
The primary objective of the study is to describe absolute lymphocyte count (ALC) reconstitution after Dimethyl fumarate (DMF) discontinuation, in Relapsing-Remitting Multiple Sclerosis (RRMS) participants with lymphopenia.

The secondary objectives of the study are characterization of lymphopenia in overall population; characterization of lymphopenia in participant with DMF discontinuation ; description of the evolution of ALC during DMF treatment; description of the time to reach a discontinuation of DMF treatment; exploration of the time to reach clinical outcomes (Expanded Disability Status Scale [EDSS] and relapse) according to lymphopenia; description of the event rate of the serious or opportunistic infections in overall population from DMF initiation and according to DMF discontinuation and lymphopenia; description of the event rate of serious and opportunistic infections in overall population from DMF initiation and according to lymphopenia; estimation of the associations between the baseline demographic and clinical characteristics and the risk to reach a lymphopenia; estimation of the associations between the baseline demographics and clinical characteristics and the risk to reach an ALC reconstitution after DMF discontinuation in participants with lymphopenia; and investigation of the changes of absolute cluster of differentiation 4 (CD4) and cluster of differentiation 8 (CD8) count in overall population on DMF if available.

DETAILED DESCRIPTION:
The study will select participants initiating treatment from 01 Jan 2016 to 15 Dec 2020.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of RRMS at DMF initiation
* Minimum of 3 months of continuous treatment with DMF*
* Initiation of DMF between January 1st, 2016 and December 15th, 2020
* Minimum of 2 ALC assessments:

  1. 1 ALC at DMF initiation (or within 6 months before DMF initiation); or under DMF treatment
  2. 1 ALC before the database extraction (15/06/2021).

     * to avoid the early DMF discontinuations for reasons other than lymphopenia.

Exclusion Criteria:

* Participants will be excluded from the study entry if they express their opposition to collect the data upon the information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All RRMS participants treated with DMF who fulfil the inclusion criteria are eligible to participate in the study.
Sampling Method: Probability Sample
Enrollment: 1507 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Time to ALC Reconstitution After DMF Discontinuation | Up to end of study (121 days)

SECONDARY OUTCOMES:
Time From DMF Initiation to Lymphopenia Initiation Assessed in Participants With and Without DMF Discontinuation | Up to end of study (121 days)
Time From DMF Initiation to Lymphopenia Assessed at Time of DMF Discontinuation | Up to end of study (121 days)
  This outcome measure will be assessed in subgroup of participants who discontinued DMF in the lymphopenic population.
Percent Change in ALC Over Time From DMF Initiation to DMF Discontinuation or End of Study | Up to end of study (121 days)
Time From DMF Initiation to DMF Discontinuation | Up to end of study (121 days)
Percentage of Participants with Discontinuation of DMF Treatment | Up to end of study (121 days)
Time to DMF Discontinuation to the First Relapses and/or an EDSS Progression | Up to end of study (121 days)
  EDSS is based on a standardized neurological exam and focuses on symptoms that commonly occur in multiple sclerosis (MS). Scores range from 0.0 (normal) to 10.0 (death due to MS).
Percentage of Participants With Serious or Opportunistic Infections in Overall and According to DMF On-going or not and in Lymphopenic Population | Up to end of study (121 days)
Percentage of Participants With Serious and Opportunistic Infections in Overall and in Lymphopenic Population | Up to end of study (121 days)
Time to Occurrence of Lymphopenia During DMF Treatment Assessed in Association Between Demographic and Clinical Characteristics | Up to end of study (121 days)
  Association between baseline demographic and clinical characteristics like age at DMF initiation, gender, diabetes, smoking habits, first ALC value close to DMF initiation, disease duration at DMF initiation, number of relapses in prior year, baseline EDSS, and any prior DMT will be assessed in this outcome measure.
Time to Lymphocyte Reconstitution After DMF Discontinuation Assessed in Association Between Demographic and Clinical Characteristics | Up to end of study (121 days)
  Association between baseline demographic and clinical characteristics like age at DMF discontinuation, gender, diabetes, smoking habits, last ALC during DMF, disease duration at DMF discontinuation, number of relapses in prior year before DMF initiation, EDSS at DMF discontinuation, DMF duration (overall, up to lymphopenia, after lymphopenia), any prior DMT, and grade of lymphopenia will be assessed in this outcome measure.
Percent Change from Baseline in Absolute CD4+ Count | Up to end of study (121 days)
Percent Change from Baseline in Absolute CD8+ Count | Up to end of study (121 days)
Percent Change from Baseline in Absolute CD4+/CD8+ Ratio | Up to end of study (121 days)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (32):
- France (32):
  - Research Site, Amiens
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Caen
  - Research Site, Clermont-Ferrand
  - Research Site, Dijon
  - Research Site, Grenoble
  - Research Site, Île-de-France - Bicêtre
  - Research Site, Île-de-France - Créteil
  - Research Site, Île-de-France - Poissy St-Germain
  - Research Site, Île-de-France - Pontoise
  - Research Site, Île-de-France - Rothschild
  - Research Site, Île-de-France - Saint-Antoine
  - Research Site, Île-de-France - Saint-Denis
  - Research Site, Île-de-France - Salpêtrière
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nancy
  - Research Site, Nantes
  - Research Site, Nice
  - Research Site, Nîmes
  - Research Site, Poitiers
  - Research Site, Rennes
  - Research Site, Rouen
  - Research Site, Saint-Etienne
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Tours

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] de Seze J, Labauge P, Liblau R, Martinez M, Moreau T, Suchet L, Vermersch P, Vukusic S, Mathey G, Michel L, Ciron J, Ruet A, Maillart E, Zephir H, Papeix C, Defer G, Cohen M, Laplaud DA, Berger E, Clavelou P, Thouvenot E, Heinzlef O, Pelletier J, Giannesini C, Casez O, Bourre B, Wahab A, Magy L, Camdessanche JP, Doghri I, Labeyrie C, Hankiewicz K, Neau JP, Pottier C, Dobay P, Li H, Levin S, Gros M, Ruiz M, Rollot F. LymphoTEC: a Retrospective Real-World Study on Lymphocyte Reconstitution After Lymphopenia in Patients with Multiple Sclerosis Treated with Dimethyl Fumarate in France. Adv Ther. 2025 Apr;42(4):1760-1782. doi: 10.1007/s12325-024-03092-5. Epub 2025 Feb 19. PMID 39969782